CLINICAL TRIAL: NCT03861793
Title: A Phase 1/2 Study of ALKS 4230 Administered Subcutaneously as Monotherapy and in Combination With Pembrolizumab in Subjects With Advanced Solid Tumors - ARTISTRY-2 (001)
Brief Title: A Dose Escalation and Cohort Expansion Study of Subcutaneously-Administered Cytokine ALKS 4230 (Nemvaleukin Alfa) as a Single Agent and in Combination With Anti-PD-1 Antibody (Pembrolizumab) in Subjects With Select Advanced or Metastatic Solid Tumors (ARTISTRY-2)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mural Oncology, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALKS 4230-001
Record Dates: First submitted 2019-02-25; First posted 2019-03-04 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Advanced Solid Tumors
Keywords: Alkermes; IL-2; Interleukin-2; Oncology; Immuno-oncology; Cytokine; ALKS 4230; Pembrolizumab; Keytruda; PD-L1; Solid tumors; Immunotherapy; nemvaleukin alfa; ovarian; Head and Neck; NSCLC; Non small cell lung cancer; lung cancer; Gastric; Gastric Cancer; Gastroesophageal Cancer; Gastroesophageal junction (GEJ) adenocarcinoma; GEJ Cancer; adenocarcinoma
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Stomach Neoplasms; Adenocarcinoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALKS 4230 (Experimental): Administered via SC injection once every 7 days or once every 21 days at escalating doses
  Interventions: Biological: ALKS 4230
- ALKS 4230 + pembrolizumab (Experimental): ALKS 4230 will be administered via SC injection once every 7 or 21 days at escalating doses or at the recommended phase 2 dose and schedule; pembrolizumab will be administered as an intravenous infusion given over 30 minutes; the dose level for pembrolizumab will be 200 mg per the approved label. In December 2020, an RP2D of 3 mg with an administration schedule of q7d was determined for SC ALKS 4230.
  Interventions: Biological: ALKS 4230; Biological: Pembrolizumab

INTERVENTIONS:
Biological: ALKS 4230 — SC injection administered in the back of the arm or the abdomen
Biological: Pembrolizumab — Administered as an intravenous (IV) infusion over 30 minutes
  Other Names: Keytruda
  Arms: ALKS 4230 + pembrolizumab

SUMMARY:
This study will characterize the safety and tolerability and identify the recommended Phase 2 dose (RP2D) of subcutaneous (SC) ALKS 4230 as monotherapy and in combination with pembrolizumab.

DETAILED DESCRIPTION:
This study will evaluate ALKS 4230 administered SC as lead-in monotherapy and in combination with pembrolizumab in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* For Phase I the subject has histological or cytological evidence of a solid tumor. For Phase II the subject must have 1 of the specified adult solid tumor types: gastric, ovarian, lung, head and neck.
* Subject must have at least one target lesion based on RECIST
* Subject has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 1
* Subjects must have adequate liver function
* Subjects must have adequate kidney function
* Subjects must be recovered from the effects of any prior chemotherapy, immunotherapy, other prior systemic anticancer therapy, radiotherapy or surgery
* Subjects who have received radiation therapy must wait at least 4 weeks after their last radiation treatment before enrollment into the study
* Females of childbearing potential must have a negative pregnancy test within 7 days of the start of treatment and on Day 1 before the first dose is administered
* Subject will agree to follow contraceptive requirements defined in the protocol
* Additional criteria may apply

Exclusion Criteria:

* Subject is currently pregnant, planning to become pregnant, or breastfeeding
* Subjects with an active infection or with a fever ≥ 38.5°C within 3 days of the first scheduled day of dosing for Cycle 1
* Subjects with active or symptomatic central nervous system metastases are excluded. Subjects with central nervous system metastases are eligible for the study if the metastases have been treated by surgery and/or radiation therapy, the subject is off corticosteroids for at least 2 weeks, and the subject is neurologically stable
* Subjects with known hypersensitivity to any components of ALKS 4230 or to pembrolizumab or any of its excipients
* Subjects who require pharmacologic doses of systemic corticosteroids are excluded; replacement doses, topical, ophthalmologic, and inhalational steroids are permitted
* Subjects who developed autoimmune disorders while on prior immunotherapy, including pneumonitis, nephritis, and/or neuropathy
* Subjects with any other concurrent uncontrolled illness, including mental illness or substance abuse, which may interfere with the ability of the subjects to cooperate and participate in the study
* The subject is known to be positive for human immunodeficiency virus (HIV), hepatitis B or C, or active tuberculosis, or has a known history of tuberculosis
* Additional criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs), and identify the RP2D of ALKS 4230 in Part A | From time of initiation of therapy until 30 days after last dose of study drug, assessed up to 24 months
  Includes AEs that are both serious and drug-related
Number of subjects experiencing AEs that are both serious and drug-related in Part B | From time of initiation of therapy until 30 days after last dose of study drug, assessed up to 24 months
  Includes AEs that are both serious and drug-related
Clinical Activity of combination treatment with ALKS 4230 and pembrolizumab in each Part B tumor type. | From time of therapy until the date of first documented tumor progression, assessed up to 24 months
  Overall Response rate (ORR) will be based on investigator review of radiographic and photographic images

SECONDARY OUTCOMES:
Proportion of subjects with objective evidence of Complete Response (CR)/immune CR (iCR) | From time of initiation of therapy until the date of first documented tumor progression, assessed up to 24 months
  Overall response rate (ORR) will be based on investigator review of radiographic or photographic images
Proportion of subjects with objective evidence of Partial Response (PR)/immune PR (iPR) | From time of initiation of therapy until the date of first documented tumor progression, assessed up to 24 months
  ORR will be based on investigator review of radiographic or photographic images
Duration of response in subjects with CR/iCR | Time from the first documentation of complete response, measured approximately every 6 weeks, to the first documentation of objective tumor progression or death due to any cause (estimated up to 24 months)
  CR/iCR duration
Duration of response in subjects with PR/iPR | Time from the first documentation of complete response, measured approximately every 6 weeks, to the first documentation of objective tumor progression or death due to any cause (estimated up to 24 months)
  PR/iPR duration
Non-progression for Part B | Assessed up to 24 months
  Time from first dose of SC ALKS 4230 to the time of progression or death
Overall survival for Part B | Assessed up to 24 months
  Time from first dose of SC ALKS 4230 to the time of death
Serum concentrations of ALKS 4230 will be determined at various time points | From time of initiation of therapy until the last treatment cycle (each cycle is 21 days), assessed up to 24 months
  Concentration vs time and standard pharmacokinetic (PK) parameters will be summarized by dose level
Serum will be assayed for the presence of anti-ALKS 4230 antibodies | From time of initiation of therapy until the last treatment cycle (each cycle is 21 days), assessed up to 24 months
  Results will be summarized by dose level
Immunophenotyping of peripheral blood mononuclear cells will be performed by flow cytometry at various time points | From time of initiation of therapy until the last treatment cycle (each cycle is 21 days), assessed up to 24 months
  Results will be summarized by dose level
Serum concentrations of proinflammatory cytokines will be assessed using a multiplex method at various time points | From time of initiation of therapy until the last treatment cycle (each cycle is 21 days), assessed up to 24 months
  Results will be summarized by dose level

CONTACTS AND LOCATIONS:
Overall Officials: Mural Oncology Medical Director, Study Director — Mural Oncology
Locations (40):
- United States (16):
  - Mural Oncology Investigational Site, Los Angeles, California
  - Mural Oncology Investigational Site, Washington D.C., District of Columbia
  - Mural Oncology Investigational Site, Atlanta, Georgia
  - Mural Oncology Investigational Site, Chicago, Illinois
  - Mural Oncology Investigational Site, Bethesda, Maryland
  - Mural Oncology Investigational Site, Detroit, Michigan
  - Mural Oncology Investigational Site, Saint Paul, Minnesota
  - Mural Oncology Investigational Site, Morristown, New Jersey
  - Mural Oncology Investigational Site, Buffalo, New York
  - Mural Oncology Investigational Site, Huntersville, North Carolina
  - Mural Oncology Investigational Site, Cincinnati, Ohio
  - Mural Oncology Investigational Site, Philadelphia, Pennsylvania
  - Mural Oncology Investigational Site, Charleston, South Carolina
  - Mural Oncology Investigational Site, Houston, Texas
  - Mural Oncology Investigational Site, Salt Lake City, Utah
  - Mural Oncology Investigational Site, Milwaukee, Wisconsin
- Canada (5):
  - Mural Oncology Investigational Site, Edmonton, Alberta
  - Mural Oncology Investigational Site, Hamilton, Ontario
  - Mural Oncology Investigational Sites, Montreal, Quebec
  - Mural Oncology Investigational Site, Montreal, Quebec
  - Mural Oncology Investigational Site, Québec, Quebec
- Netherlands (2):
  - Mural Oncology Investigational Site, Rotterdam
  - Mural Oncology Investigational Site, Utrecht
- South Korea (8):
  - National Cancer Center, Goyang
  - Inha University Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea St. Vincent's Hospital, Suwon
- Spain (5):
  - Mural Oncology Investigational Site, Badalona
  - Mural Oncology Investigational Site, Córdoba
  - Mural Oncology Investigational Site, Madrid
  - Mural Oncology Investigational Site, Málaga
  - Mural Oncology Investigational Site, Valencia
- Taiwan (4):
  - Mural Oncology Investigational Site, Kaohsiung City
  - Mural Oncology Investigational Site, Taichung
  - Mural Oncology Investigational Site, Tainan
  - Mural Oncology Investigational Site, Taipei

IPD SHARING:
Plan to Share IPD: No
At this time, IPD sharing has not been defined and/or decided if it will be shared.